CLINICAL TRIAL: NCT01735058
Title: Evaluating the Efficacy of Ultrasonography Guided Subacromial Sodium Hyaluronate Injection in the Treatment of Rotator Cuff Disease
Brief Title: Ultrasonography Guided Subacromial Sodium Hyaluronate Injection in Rotator Cuff Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Farnaz Dehgan Hosseinabadi, Principal Investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13912134
Record Dates: First submitted 2012-11-16; First posted 2012-11-28 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Hyaluronic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium hyaluronate (Active Comparator): Ultrasound guided injection of sodium hyaluronate
  Interventions: Drug: Sodium Hyaluronate
- Normal saline (Placebo Comparator): Ultrasound guided injection of normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Sodium Hyaluronate — Ultrasound guided injection of sodium hyaluronate; Fermathron ™, 20 mg/2ml of Sodium Hyaluronate, 3 weekly injections.
  Arms: Sodium hyaluronate
Drug: Normal saline — Ultrasound guided injection of 0.9% normal sodium hyaluronate line solution, at 2 mL/syringe, 3 weekly injections.
  Arms: Normal saline

SUMMARY:
This study will be performed to examine the effect of ultrasound-guided subacromial sodium hyaluronate injection in patients with impingement syndrome without rotator cuff complete tear.

DETAILED DESCRIPTION:
Rotator cuff disease in particular is a common cause of shoulder pain and weakness and comprises a significant proportion of the musculoskeletal complaints presenting to primary care doctors. Ultrasound is a readily available and cheap modality for looking more specifically at the rotator cuff and surrounding structures. More recently, ultrasound guidance has become a commonly employed method to perform diagnostic or therapeutic interventions. Despite the long history and the fact that this is a common diagnosis made in clinical practice, the exact cause and best treatment for this condition still are being explored. Although there are a few high-quality studies demonstrating the efficacy of sodium hyaluronate injection for rotator cuff disease, this study will be performed to examine the effect of ultrasound-guided subacromial sodium hyaluronate injection in patients with impingement syndrome without rotator cuff complete tear.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* subacromial impingement syndrome
* without a complete tear of rotator cuff
* willingness to participate

Exclusion Criteria:

* had any rheumatic disease, glenohumeral osteoarthritis, full-thickness rotator cuff tears, fractures, diabetes mellitus, infections, or tumors.
* had hypersensitivity to hyaluronate
* had participated in any other study within 6 months
* had received a subacromial injection within 8 weeks
* were pregnant or planned to become pregnant
* were at risk of complications of intra-articular injections such as patients who received anti-coagulant drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain severity after 3 weeks. | Up to 3 weeks
  The pain score (100 mm Visual Analogue Score ) is evaluated before the first injection and one week after each injection up to 3rd week.

CONTACTS AND LOCATIONS:
Overall Officials: Farnaz Dehghan, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Department of Rehabilitation, Alzahra Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Andrews JR. Diagnosis and treatment of chronic painful shoulder: review of nonsurgical interventions. Arthroscopy. 2005 Mar;21(3):333-47. doi: 10.1016/j.arthro.2004.11.003. PMID 15756189
- [Background] Meloni F, Milia F, Cavazzuti M, Doria C, Lisai P, Profili S, Meloni GB. Clinical evaluation of sodium hyaluronate in the treatment of patients with sopraspinatus tendinosis under echographic guide: experimental study of periarticular injections. Eur J Radiol. 2008 Oct;68(1):170-3. doi: 10.1016/j.ejrad.2007.11.001. Epub 2007 Dec 21. PMID 18096343
- [Background] Kim YS, Park JY, Lee CS, Lee SJ. Does hyaluronate injection work in shoulder disease in early stage? A multicenter, randomized, single blind and open comparative clinical study. J Shoulder Elbow Surg. 2012 Jun;21(6):722-7. doi: 10.1016/j.jse.2011.11.009. Epub 2012 Feb 25. PMID 22366365
- [Background] Chou WY, Ko JY, Wang FS, Huang CC, Wong T, Wang CJ, Chang HE. Effect of sodium hyaluronate treatment on rotator cuff lesions without complete tears: a randomized, double-blind, placebo-controlled study. J Shoulder Elbow Surg. 2010 Jun;19(4):557-63. doi: 10.1016/j.jse.2009.08.006. Epub 2009 Dec 5. PMID 19963403